CLINICAL TRIAL: NCT06975644
Title: A Prospective Clinical Study Evaluating Bemotuzumab Combined With Chemotherapy to Improve the Efficacy of Neoadjuvant Chemotherapy for Triple-Negative Breast Cancer (TNBC)
Brief Title: Evaluating Bemotuzumab to Improve the Efficacy of Neoadjuvant Chemotherapy for Triple-Negative Breast Cancer (TNBC)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhejiang Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Xuli Meng, Chief physician, Zhejiang Provincial People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LuxMed 01
Record Dates: First submitted 2025-05-09; First posted 2025-05-16 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-04

CONDITIONS: Triple-Negative Breast Cancer (TNBC); Neoadjuvant Chemotherapy; Chemotherapy Effects
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — 130-nm albumin-bound paclitaxel; Carboplatin; Epirubicin; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single-Arm Trial (Experimental): Patients meeting the eligibility criteria will receive neoadjuvant chemotherapy combined with immunotherapy: 4 cycles of nab-paclitaxel, carboplatin, and bemotuzumab, followed by 4 cycles of epirubicin, cyclophosphamide, and bemotuzumab
  Interventions: Drug: nab-paclitaxel, carboplatin, and bemotuzumab; Drug: epirubicin, cyclophosphamide, and bemotuzumab

INTERVENTIONS:
Drug: nab-paclitaxel, carboplatin, and bemotuzumab — nab-paclitaxel：260 mg/m2 Q3W；carboplatin：AUC 6；bemotuzumab：1200 mg Q3W
Drug: epirubicin, cyclophosphamide, and bemotuzumab — epirubicin：90 mg/m2 Q3W；cyclophosphamide：600 mg/m2 Q3W；bemotuzumab：1200 mg Q3W

SUMMARY:
Evaluating Bemotuzumab to improve the efficacy of neoadjuvant chemotherapy for Triple-Negative Breast Cancer (TNBC)

DETAILED DESCRIPTION:
This study aims to prospectively evaluate the pathological complete response (pCR) rate in patients with early-stage triple-negative breast cancer (TNBC) receiving standard neoadjuvant chemotherapy combined with bemotuzumab.

ELIGIBILITY:
Inclusion Criteria:

* 1.Voluntarily agree to participate in the clinical study and sign the informed consent form.
* 2.Female patients aged ≥18 years at the time of signing the informed consent form.
* 3.Women of childbearing potential (WOCBP) must have a negative serum pregnancy test within 7 days prior to enrollment and agree to use a clinically recognized highly effective contraceptive method during the study and for 3 months after the last dose of the study drug.
* 4.Adequate archival tumor tissue samples for HIM-type analysis (at least 15 unstained tumor biopsy slides from the most recent metastatic lesion; archival primary tumor samples from treatment-naïve patients are acceptable, or re-biopsied specimens may be submitted).
* 5.Primary breast cancer meeting the following criteria:Histologically confirmed invasive breast cancer.Breast cancer staging (AJCC 8th edition): T1c-4, N0-2, M0.Histopathologically confirmed triple-negative invasive breast cancer (TNBC) meeting all criteria:HER2-negative: IHC 0/1+ or IHC 2+ with negative in situ hybridization (ISH).ER-negative: IHC <1%.PR-negative: IHC <1%.Unstained tumor sections must be submitted to the central laboratory as per the study protocol for biomarker validation.
* 6.Willingness to undergo surgery if deemed eligible after neoadjuvant therapy.
* 7.Adequate organ function as defined by protocol-specified laboratory thresholds.
* 8.Eastern Cooperative Oncology Group (ECOG) performance status score ≤1 within 7 days prior to the first dose.

Exclusion Criteria:

* 1. Pathological Staging a) Inflammatory breast cancer.b) Stage IV (metastatic) breast cancer, bilateral breast cancer, or multicentric breast cancer (defined as multifocal tumors involving more than one quadrant with lesions separated by ≥5 cm).
* 2. Tumor-Related Conditions a) Radiologic evidence of tumor invasion into major blood vessels or investigator-determined high risk of life-threatening hemorrhage due to impending vascular compromise.b) Uncontrolled or symptomatic hypercalcemia (>1.5 mmol/L ionized calcium, >12 mg/dL serum calcium, or albumin-corrected serum calcium > upper limit of normal [ULN]); or symptomatic hypercalcemia requiring ongoing bisphosphonate therapy.c) Other severe concurrent illnesses interfering with treatment plans, including significant pulmonary conditions/diseases.
* 3. Prior/Concurrent Anticancer Therapies a) Previous or current systemic antitumor therapy for the current breast cancer (including chemotherapy, molecular targeted therapy, biologic therapy, or investigational agents).b) Participation in another clinical trial within 4 weeks prior to enrollment (3 months for monoclonal antibody trials) or planned participation during this study.c) Prior treatment with immune checkpoint inhibitors other than PD-1/PD-L1 monoclonal antibodies (e.g., CTLA-4 inhibitors) or anti-angiogenic agents (including monoclonal antibodies or TKIs).d) Administration of live/attenuated vaccines within 28 days before the first dose or anticipated vaccination during the study.
* 4. Medical History/Comorbidities a) Other malignancies within the past 5 years requiring systemic/local therapy (excluding cured carcinoma in situ, cervical intraepithelial neoplasia, basal/squamous skin cancer, or thyroid cancer).b) Major surgery within 28 days before the first dose (defined as requiring ≥3 weeks recovery) or palliative radiotherapy/ablation within 2 weeks.c) Known/suspected autoimmune diseases, except:Hypothyroidism managed with hormone replacement.Stable type 1 diabetes with controlled glycemia.d) Active viral hepatitis:HBV: HBsAg(+) or HBcAb(+) with HBV-DNA(+) (except those with HBV-DNA ≤2,500 copies/mL or 500 IU/mL after antiviral therapy).HCV: HCV-Ab(+) with HCV-RNA(+).Coinfection with HBV and HCV.e) HIV infection (HIV-Ab(+)).f) Interstitial lung disease, non-infectious pneumonitis, or uncontrolled systemic diseases (e.g., diabetes, pulmonary fibrosis, acute pneumonitis).g) Severe infections:Hospital-required infections (e.g., bacteremia, pneumonia) within 4 weeks.Active CTCAE ≥Grade 2 infections requiring systemic antibiotics within 2 weeks.Unexplained fever >38.5°C during screening (tumor-related fever permitted per investigator).Active tuberculosis within 1 year.h) Prior allogeneic bone marrow or solid organ transplantation.i) Peripheral neuropathy ≥Grade 2 (CTCAE v5.0).j) History of neurological/psychiatric disorders (e.g., epilepsy, dementia), drug/alcohol abuse.k) Significant cardiac disease:Heart failure (LVEF <50%).High-risk arrhythmias (resting HR >100 bpm, ventricular tachycardia, Mobitz II/third-degree AV block).Unstable angina requiring antianginal therapy.Clinically significant valvular disease.ECG-confirmed transmural myocardial infarction.Uncontrolled hypertension (systolic >180 mmHg/diastolic >100 mmHg).
* 5. Treatment-Related Exclusions a) Systemic immunostimulants (e.g., interferon, interleukin-2) within 4 weeks before the first dose.b) Systemic immunosuppressants (e.g., glucocorticoids, azathioprine) within 2 weeks, except:Topical/inhaled corticosteroids.Physiologic steroid replacement (≤10 mg/day prednisone equivalent).c) Hypersensitivity to study drug components or severe allergic reactions to monoclonal antibodies.
* 6. Pregnancy/Lactation Pregnant/lactating women or women of childbearing potential with positive baseline pregnancy tests or unwilling to use effective contraception.
* 7. Investigator Discretion Any condition deemed by the investigator to compromise protocol compliance or patient safety.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response | six months

CONTACTS AND LOCATIONS:
Overall Officials: Xuli Meng, Study Chair — Zhejiang Provincial People's Hospital

IPD SHARING:
Plan to Share IPD: No
After preliminary results are available, it is advisable to decide whether to share them with other researchers.